CLINICAL TRIAL: NCT00006467
Title: Phase II Trial of Gemcitabine and ISIS 2503 in Patients With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Gemcitabine and ISIS 2503 in Treating Patients With Advanced or Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0043; CDR0000068281 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-11-06; First posted 2004-03-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; duct cell adenocarcinoma of the pancreas; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ISIS 2503; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + ISIS 2503 (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and ISIS 2503 IV continuously on days 1-14. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: ISIS 2503; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: ISIS 2503
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with ISIS 2503 in treating patients who have advanced or metastatic cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the 6-month and overall survival rates in patients with locally advanced or metastatic adenocarcinoma of the pancreas treated with gemcitabine and ISIS 2503. II. Determine the response rate of these patients treated with this regimen. III. Assess the toxicity of this regimen in this patient population.

OUTLINE: This is a multicenter study. Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and ISIS 2503 IV continuously on days 1-14. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally advanced or metastatic adenocarcinoma of the pancreas not amenable to standard curative therapy Duct cell Undifferentiated The following cellular types are not eligible: Islet cell carcinoma Acinar cell carcinoma Cystadenocarcinoma No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 No underlying disease associated with active bleeding Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN AST no greater than 3 times ULN PT and PTT normal Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy or immunotherapy No concurrent immunotherapy No colony-stimulating factors during first course of therapy Chemotherapy: No prior chemotherapy except radiosensitizing agents used in adjuvant setting or in treatment of locally advanced disease No prior gemcitabine No prior ISIS 2503 No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to 25% or greater of bone marrow No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-02; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
overall survival at 6 months | at 6 months

SECONDARY OUTCOMES:
response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Alberts SR, Schroeder M, Erlichman C, Steen PD, Foster NR, Moore DF Jr, Rowland KM Jr, Nair S, Tschetter LK, Fitch TR. Gemcitabine and ISIS-2503 for patients with locally advanced or metastatic pancreatic adenocarcinoma: a North Central Cancer Treatment Group phase II trial. J Clin Oncol. 2004 Dec 15;22(24):4944-50. doi: 10.1200/JCO.2004.05.034. PMID 15611509